CLINICAL TRIAL: NCT04449510
Title: Short-Term Cardiovascular Effects of E-Cigarettes: Influence of E-Liquid pH
Acronym: TCORS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-30597; 5U54HL147127-09 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Risk Factor; Nicotine Dependence
Keywords: E-Cigarettes; Vaping; E-Cig Mods
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-liquid pH 5, 7, or 9 (Other): Using an electronic cigarette, the participant will complete a standardized vaping session using 1 of 3 assigned e-liquid pH.
  Interventions: Other: Electronic Cigarette
- 1 of the other 2 remaining e-liquid pH (Other): Using an electronic cigarette, the participant will complete a standardized vaping session using 1 of the other 2 assigned e-liquid pH.
  Interventions: Other: Electronic Cigarette
- Remaining e-liquid pH (Other): Using an electronic cigarette, the participant will complete a standardized vaping session using the remaining assigned e-liquid pH.
  Interventions: Other: Electronic Cigarette

INTERVENTIONS:
Other: Electronic Cigarette — E-cigarette Device: The delivery device will be a variable wattage all-in-one device with operating wattage of 7.0 - 75.0 W. The device will be set at 10 watts for the study visits.

SUMMARY:
This study will examine the short-term cardiovascular (CV) effects of e-liquid pH in a randomized, crossover clinical and behavioral pharmacology study of experienced adult e-cigarette users (N=21). The specific aim is to determine the impact of e-cigarette pH levels on nicotine pharmacology, systemic exposure to toxic volatile organic compounds (VOCs), and short-term cardiovascular effects.

DETAILED DESCRIPTION:
This is a single-site, randomized, crossover study of experienced adult e-cigarette users to assess nicotine exposure, toxicant exposure, and the short-term CV effects of e-liquid pH. Three e-liquid pH conditions will be assessed on all participants: 5, 7, and 9.

Hypothesis 2a: The rate of systemic nicotine absorption is inversely related to e-liquid pH and results in lower peak blood nicotine levels at higher pH.

Hypothesis 2b: Heart rate acceleration will decrease and subjective measures of sensation in the throat, reward, and satisfaction will increase with increasing e-liquid pH.

ELIGIBILITY:
Inclusion Criteria:

* Heart rate < 105 beats per minute (BPM)*
* Systolic Blood pressure <160 and > 90*
* Diastolic Blood Pressure <100 and > 50*
* Body Mass Index (BMI) < 38.0 (at investigator's discretion for higher BMI if no other concurrent health issues)

  *considered out of range if both machine and manual readings are above/below these thresholds
* Use e-cigarettes on at least 15 days in the past 30 for at least 3 months
* Smoke 10 or fewer cigarettes/tobacco products per day in the last 30 days
* Willing to use mod e-cigarette
* Willing to abstain from tobacco product use for night before study
* Age: > 21 years old and < 70 years old
* Using e-liquid > 0mg/ml nicotine
* Saliva cotinine of ≥ 30 ng/ml or NicAlert=6 (in cases where lab turn around time will delay study procedure)

Exclusion Criteria:

* Seizures
* Cancer
* Hepatitis B or C or Liver Disease
* Oral Thrush
* Heart disease
* Glaucoma
* Kidney disease or urinary retention
* Diabetes
* High Blood Pressure (taking sympatholytic medications such as alpha and beta blockers)
* History of stroke
* An ulcer in the past year
* Thyroid disease (okay if controlled with medication)
* Active use of an inhaler for asthma or Chronic Obstructive Pulmonary Disease (COPD)
* Psychiatric conditions
* Current or past schizophrenia, and/or current or past bipolar disorder
* Major depression, current or within the past year
* Major personality disorder
* Participants with current or past minor or moderate depression and/or anxiety disorders will be reviewed by the study physician and considered for inclusion.
* History of psychiatric hospitalizations are not exclusionary, but study participation will be determined as per study physician's approval
* Recent onset or change in cough, fever and/or abdominal symptoms (vomiting or pain) in the past two weeks. (If yes, participant can re-screen when symptoms resolve).
* Drug/Alcohol Dependence
* Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program
* Positive toxicology test at the screening visit (THC & prescribed medications okay)
* Opioid replacement therapy (including methadone, buprenorphine, or other)
* Positive urine cannabis is not exclusionary but participant must report use of cannabis and agree to abstain from cannabis use for the duration of the study
* Psychiatric medications
* Current regular use of any psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitor (SSRI) and serotonin-norepinephrine reuptake Inhibitor (SNRIs) and current evaluation by the study physician that the participant is otherwise healthy, stable, and able to participate.
* Medications
* Use of medications that are inducers of nicotine metabolizing enzyme CYP2A4 (Example: rifampicin, carbamazepine, phenobarbital, and other anticonvulsant drugs).
* Concurrent use of nicotine-containing medications
* Any stimulant medications (example: Adderall) generally given for Attention deficit hyperactivity disorder (ADHD) treatment
* Use of sympatholytic medications that affect cardiovascular conditions including hypertension, (Example: beta and alpha-blockers)
* Other/Misc. Chronic Health Conditions
* Fainting (within the last 30 days)
* Other "life threatening illnesses" as per study physician's discretion
* Pregnancy
* Pregnancy (self-reported and urine pregnancy test)
* Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial
* Inability to communicate in English
* Planning to quit vaping within the next 60 days
* Uncomfortable with getting blood drawn

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Mean Blood Nicotine Level | Day 1 of each Arm
  Concentration of plasma nicotine (ng/ml) will be used to assess differences across the three e-liquid pH levels.
Mean Saliva pH | Day 1 of each Arm
  Participant saliva pH will be measured before and during outpatient stay.
Mean Heart Rate | Day 1 of each Arm
  Participant heart rate will be measured in beats per minute throughout the outpatient stay.
Mean Skin Blood Flow | Day 1 of each Arm
  Participant skin blood flow will be measured by product of average blood cell velocity and concentration in mL/min during outpatient stay.
Mean scores on the Minnesota Nicotine Withdrawal Scale (MNWS) | Day 1 of each Arm
  The investigators will compile a score for the subjective effect of withdrawal using the sum of points scored on the Minnesota Nicotine Withdrawal Scale (MNWS), where a higher score (score range from 0 points to 60 points) indicates a higher intensity of the indicated subjective effect.
Mean scores on the Questionnaire of Smoking Urges (QSU-Brief) | Day 1 of each Arm
  The investigators will compile a score for the subjective effect of craving using the sum of points scored in the two subscales (intention and desire to engage in smoking behavior that is anticipated as pleasant, and anticipation of relief from negative affect through smoking) of the Questionnaire of Smoking Urges (QSU-Brief), where a higher score (score range from 10 points to 70 points) indicates a higher intensity of the indicated subjective effect.
Mean scores on the Cigarette Evaluation Scale (mCES) | Day 1 of each Arm
  The investigators will compile a score for the subjective effect of reward using the sum of points scored in the five subscales (Smoking Satisfaction - score range from 1 point to 7 points; Psychological Reward - score range from 5 points to 35 points; Aversion - score range from 2 points to 14 points; Enjoyment of Respiratory Tract Sensations - score range from 2 points to 14 points; and Craving Reduction - score range from 1 point to 7 points) of the modified Cigarette Evaluation Scale (mCES), where a higher score indicates a higher intensity of the indicated subjective effect.

SECONDARY OUTCOMES:
Mean puffs per minute | Day 1 of each Arm
  Vaping topography measures will be obtained from frame by frame analysis of high definition videos during the ad libitum sessions and measured as puffs per minute.
Mean seconds per puff | Day 1 of each Arm
  Vaping topography measures will be obtained from frame by frame analysis of high definition videos during the ad libitum sessions and measured as seconds per puff.
Mean time between puffs | Day 1 of each Arm
  Vaping topography measures will be obtained from frame by frame analysis of high definition videos during the ad libitum sessions and measured as seconds/minutes between puffs.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon St. Helen, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with research collaborators during the course of the study.

DOCUMENTS (1):
  • Informed Consent Form (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04449510/ICF_000.pdf